CLINICAL TRIAL: NCT01148771
Title: Comparative Pharmacokinetics, Safety, and Pharmacodynamics of Ertapenem 1 Gram Daily Administered as an IV Bolus Versus Standard 30 Minute Infusion to Healthy Adult Volunteers
Brief Title: Pharmacokinetics (PK) of Ertapenem Intravenous (IV) Bolus Versus Standard Infusion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hartford Hospital (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: KUTI003194HE; IISP ID#37935 (Other Grant/Funding Number: Merck)
Record Dates: First submitted 2010-06-18; First posted 2010-06-22 (Estimated); Results first posted 2012-05-11 (Estimated); Last update posted 2012-05-11 (Estimated); Status verified 2012-04

CONDITIONS: Healthy
Keywords: Pharmacokinetics; Safety
MeSH Terms: interventions — Ertapenem

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ertapenem 1 gram intravenous (IV) 5 minute bolus (Experimental): Participants received ertapenem 1 gram every 24 hours for 3 doses with each dose infused as a 5 minute IV bolus.
  Interventions: Drug: ertapenem
- Ertapenem 1 gram IV 30 minute infusion (Active Comparator): Participants received ertapenem 1 gram every 24 hours for 3 doses with each dose infused as a 30 minute infusion (i.e., the standard dose).
  Interventions: Drug: ertapenem

INTERVENTIONS:
Drug: ertapenem — 1 gram IV bolus every 24 hours (q24h) for 3 days
  Arms: Ertapenem 1 gram intravenous (IV) 5 minute bolus
Drug: ertapenem — 1 gram 30 minute infusion q24h for 3 days
  Arms: Ertapenem 1 gram IV 30 minute infusion

SUMMARY:
The purpose of this study is to characterize and compare the concentration-time profiles and multiple dose pharmacokinetics of a 5 minute intravenous (IV) bolus of ertapenem 1 gram daily versus the standard 30 minute infusion in healthy volunteers. Safety and tolerability and pharmacodynamic target attainment using Monte Carlo simulation will also be assessed and compared.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults (18 years of age or older)

Exclusion Criteria:

* Ertapenem or other beta-lactam allergy
* Pregnant or breast feeding females
* Body Mass Index (BMI) greater than or equal to 30
* Abnormal lab values at baseline
* Hypertension
* Significant medical abnormality
* Regular alcohol consumption
* Significant nicotine use

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-08; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Josepth L Kuti, PharmD, Principal Investigator — Hartford Hospital; Dora E Wiskirchen, PharmD, Study Director — Hartford Hospital
Locations (1):
- Hartford Hospital, Hartford, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy adult volunteers were recruited in August/September 2010.
Pre-assignment Details: The target enrollment of 12 volunteers was met. All 12 participants completed at least one phase of the study, while 11 completed the entire study.
Groups:
- Ertapenem IV 5 Minute Bolus First, Then 30 Minute Infusion: Participants received ertapenem 1 gram as a 5 minute IV bolus every 24 hours for 3 doses. After a 4 day washout, participants were crossed over to receive ertapenem 1 gram as a 30 minute IV infusion every 24 hours for 3 doses.
- Ertapenem IV 30 Minute Infusion First, Then 5 Minute Bolus: Participants received ertapenem 1 gram as a 30 minute infusion every 24 hours for 3 doses. After a 4 day washout, participants crossed over to receive ertapenem 1 gram as a 5 minute IV bolus every 24 hours for 3 doses.
Period: First Intervention
Arm/Group | Ertapenem IV 5 Minute Bolus First, Then 30 Minute Infusion | Ertapenem IV 30 Minute Infusion First, Then 5 Minute Bolus
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0
Period: Washout Period
Arm/Group | Ertapenem IV 5 Minute Bolus First, Then 30 Minute Infusion | Ertapenem IV 30 Minute Infusion First, Then 5 Minute Bolus
Started | 6 | 6
Completed | 6 | 5
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Second Intervention
Arm/Group | Ertapenem IV 5 Minute Bolus First, Then 30 Minute Infusion | Ertapenem IV 30 Minute Infusion First, Then 5 Minute Bolus
Started | 6 | 5
Completed | 6 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ertapenem IV 5 Minute Bolus First, Then 30 Minute Infusion | Ertapenem IV 30 Minute Infusion First, Then 5 Minute Bolus | Total
Number analyzed (Participants) | 11 | 12 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 12 | 23
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 32.4 (13.9) | 32.4 (13.9) | 32.4 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 8 | 8 | 16
Region of Enrollment [Number; unit: participants]
  United States | 11 | 12 | 23

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) at Steady-State (After 3rd Dose)
Description: Cmax is measured at 5 minutes after the beginning of the infusion for the 5 minute IV bolus dosage regimen and at 30 minutes after the beginning of the infusion for the 30 minute infusion dosage regimen.
Time Frame: 5 or 30 minutes post start of infusion on Day 3
Population: Each participant received ertapenem as a 5 minute infusion and as a 30 minute infusion, only in different order due to cross-over design. Data for all participants receiving each dosage regimen are included in each arm for results.
Measure: Mean (Standard Deviation); unit: mcg/mL
Groups:
- Ertapenem 1 Gram IV 5 Minute Bolus: Participants received ertapenem 1 gram as a 5 minute IV bolus every 24 hours for 3 doses.
- Ertapenem 1 Gram IV 30 Minute Infusion: Participants received ertapenem 1 gram as a 30 minute infusion every 24 hours for 3 doses.
Arm/Group | Ertapenem 1 Gram IV 5 Minute Bolus | Ertapenem 1 Gram IV 30 Minute Infusion
Number analyzed (Participants) | 11 | 12
mcg/mL | 193.33 (43.27) | 165.70 (20.38)

2. Secondary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability
Description: The following laboratory assessments will be make before and after participation in the study to determine if objective changes occurred: blood pressure, pulse rate, temperature, complete blood count with differential, platelet count, blood urea nitrogen, serum creatinine, liver function panel [aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase], total bilirubin, and urinalysis with microscopy. Monitoring of other pathologic or unintended changes in structure (signs),or function (symptoms) of the body associated with participation in the study will occur.
Time Frame: 3 days
Measure: Number; unit: participants
Arm/Group | Ertapenem IV 5 Minute Bolus | Ertapenem IV 30 Minute Infusion
Number analyzed (Participants) | 11 | 12
participants | 10 | 9

3. Secondary Outcome: Probability of Target Attainment (PTA)
Description: After simulating 5000 patients receiving each dosing regimen, the probability of achieving free drug concentrations above an MIC of 0.25 mcg/mL and 0.5mcg/mL for at least 40% of the dosing interval (40% fT>MIC) is calculated at each MIC dilution.
Time Frame: Simulated Steady-State Exposure
Population: The probability of achieving 40% T>MIC is reported at a MIC of 0.25mcg/mL and 0.5mcg/mL respectively.
Measure: Number; unit: % of 5000 simulated patients
Units Other Than Participants: Simulated Patients
Groups:
- Ertapenem 1 Gram IV 5 Minute Bolus: This is a simulated population of 5000 patients receiving ertapenem 1 gram every 24 hours as a 5 minute IV bolus.
- Ertapenem 1 Gram IV 30 Minute Infusion: This is a simulated population of 5000 patients receiving ertapenem 1 gram every 24 hours as a 30 minute IV infusion.
Arm/Group | Ertapenem 1 Gram IV 5 Minute Bolus | Ertapenem 1 Gram IV 30 Minute Infusion
Number analyzed (Participants) | 11 | 12
Number analyzed (Simulated Patients) | 5000 | 5000
% of 5000 simulated patients
  PTA at 0.25 | 97.0 | 97.9
  PTA at 0.5 | 1.7 | 2.8

4. Primary Outcome: Area Under the Curve From 48 to 72 Hours [AUC(48-72)]
Description: AUC(48-72) is the 24 hour area under the concentration versus time curve after the 3rd dose of ertapenem, which is selected to measure approximate AUC at steady-state.
Time Frame: 0-24 hours after 3rd ertapenem dose
Measure: Mean (Standard Deviation); unit: mcg*hr/mL
Arm/Group | Ertapenem 1 Gram IV 5 Minute Bolus | Ertapenem 1 Gram IV 30 Minute Infusion
Number analyzed (Participants) | 11 | 12
mcg*hr/mL | 561.17 (77.01) | 531.32 (56.86)

ADVERSE EVENTS:
Arm/Group | Ertapenem IV 5 Minute Bolus First, Then 30 Minute Infusion | Ertapenem IV 30 Minute Infusion First, Then 5 Minute Bolus
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/12
Other Adverse Events (participants affected / at risk) | 10/11 | 9/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ertapenem IV 5 Minute Bolus First, Then 30 Minute Infusion (N=11) | Ertapenem IV 30 Minute Infusion First, Then 5 Minute Bolus (N=12)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Headache (General disorders) | 3 (5) | 3 (7)
Diarrhea (Gastrointestinal disorders) | 6 (9) | 3 (8)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) — Reduction in Hemoglobin below normal.
Liver Function Test out of range (Hepatobiliary disorders) | 1 (1) | 2 (2) — Increases in ALT

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less